CLINICAL TRIAL: NCT04982146
Title: Intratumoral Bromelain + N-acetylcysteine in Relapsed and Unresectable Pseudomyxoma Peritonei. Phase I Single-arm Trial
Brief Title: Intratumoral Bromelain + Acetylcysteine in Relapsed and Unresectable Pseudomyxoma Peritonei
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BROAC-PMP
Record Dates: First submitted 2021-07-06; First posted 2021-07-29 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Pseudomyxoma Peritonei
Keywords: pseudomyxoma peritonei; n-acetylcysteine; acetylcysteine; NAC; bromelain
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — Bromelains; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Single-arm experimental analytical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bromelain + N-Acetylcysteine (Experimental): Patients with pseudomyxoma peritonei that are not candidates to surgical resection
  Interventions: Drug: Bromelin; Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: Bromelin — 0.5mg per mL of total tumor volume calculated, administered percutaneously
Drug: N-Acetylcysteine — 20mg per mL of total tumor volume calculated, administered percutaneously

SUMMARY:
This trial pursues studying a compassionate treatment option for patients with inoperable pseudomyxoma peritonei through percutaneous administration of bromelain + N-acetylcysteine (NAC) in order to decrease tumoral volume. Secondary endpoints are the decrease of ascites, compressive symptoms and pain through the dilution of mucins, which would better intestinal blockage.

ELIGIBILITY:
Inclusion Criteria:

* Pseudomyxoma peritonei diagnosis through imaging tests and/or histological studies
* Pseudomyxoma peritonei relapse in abdominal area in patients who comply inoperability criteria, which are:

At least two HIPEC operations or major abdominal surgery (PSS > 3). Patients with acute morbidities (ASA score IV)

* ECOG 0-2
* Age ≥ 18
* Signs informed consent

Exclusion Criteria:

* Candidates to other potentially healing treatments
* Allergy to bromelains (pineapple), N-Acetylcysteine or possible cross-reactive allergy (eggs, sulphate. latex, carrots, celery, wheat...)
* Non-manageable coagulation alterations
* No possibility of intraabdominal drainage catheter
* Acute respiratory pathology (asthma, COPD), acute hepatic, cardiopathic or kidney pathology
* Allergy to any substance that might cause crossed reactivity to bromelain
* Unwillingness to participate in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2023-05-16 (Estimated)

PRIMARY OUTCOMES:
Tumoral Mass Change | Day 3, Day 7 (if it applies),1 month and 12 months after treatment is finished.
  Tumoral mass change calculated through CT Scan or Magnetic Resonance categorized regarding the biggest diameter per abdominal region

SECONDARY OUTCOMES:
Symptoms improvement | Basal visit, 1 month and 12 months after treatment.
  Symptoms progression evaluated through QLQ-C30 questionnaire (life quality questionnaire)
TTP (Time to tumor progression) | Period of 12 months after treatment.
  Period of time free of tumor progression.
Overall survival | Period of 12 months after treatment.
  Time until death from any cause
Tumoral DNA diminution in biological samples | Basal visit, all treatment visits and 12 months after treatment is finished.
  Diminution of tumoral DNA amount found in mucin and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Rodríguez Ortiz, MD, Principal Investigator — Hospital Universitario Reina Sofía; Álvaro Arjona Sánchez, PhD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the study concludes and results are published
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After results publication
Access Criteria: Upon request to study's principal investigator